CLINICAL TRIAL: NCT03311269
Title: A Prospective, Randomized, Controlled, Multi-Center, Double Blind Study of ClariVein RES for Treatment of Venous Insufficiency Associated With Incompetent Saphenous Veins Due to Superficial Venous Reflux
Brief Title: A Study Evaluating ClariVein With a Sclerosing Agent for the Treatment of Venous Insufficiency
Acronym: VICARES
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated for administrative reasons
Sponsor: Vascular Insights, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-001
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — Sodium Tetradecyl Sulfate; Injections; 3-methoxy-14,15-methyleneestra-1,3,5-triene-17-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- ClariVein RES 1% Injection (Active Comparator): Sodium Tetradecyl Sulfate 1% Injection single administration
  Interventions: Device: ClariVein RES; Drug: Sodium Tetradecyl Sulfate 1% Injection
- ClariVein RES 3% Injection (Active Comparator): Sodium Tetradecyl Sulfate 3% Injection single administration
  Interventions: Device: ClariVein RES; Drug: Sodium Tetradecyl Sulfate 3% Injection

INTERVENTIONS:
Device: ClariVein RES — ClariVein system
Drug: Sodium Tetradecyl Sulfate 1% Injection — Sodium Tetradecyl Sulfate STS 1% Injection
  Other Names: STS 1%
  Arms: ClariVein RES 1% Injection
Drug: Sodium Tetradecyl Sulfate 3% Injection — Sodium Tetradecyl Sulfate 3% Injection
  Other Names: STS 3%
  Arms: ClariVein RES 3% Injection

SUMMARY:
VICARES is a prospective randomized, controlled, multi-center, double blind study treating venous insufficiency associated with incompetent saphenous veins with 1% and 3% Sodium Tetradecyl Sulfate (STS) solution utilizing the ClariVein system.

DETAILED DESCRIPTION:
Approximately 50 subjects diagnosed with an incompetent saphenous vein will be randomized to either 1% STS or 3% STS solution delivered by the ClariVein system under ultrasound guidance.

Study duration for individual study patients, including follow-up visits, is anticipated to be approximately 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient with incompetent saphenous vein
2. Saphenous vein reflux > 500ms (0.5s), as measured by duplex ultrasound
3. One or more of patient reported symptoms related to the target vein: i.e., heaviness, achiness, swelling, throbbing or itching.
4. Candidate for endovenous procedure

Exclusion Criteria:

1. Arterial insufficiency demonstrated by a history of peripheral arterial disease (PAD) that would preclude the wearing of compression stockings
2. Absence of a palpable pulse at posterior tibial or dorsalis pedis and an Ankle-Brachial Index (ABI) <0.6
3. Multi-segmental axial deep venous reflux in at least two contiguous venous segments (e.g., femoral and popliteal) in the ipsilateral extremity
4. Previous surgical or endovenous procedure in the treatment section of the target vein
5. Previous superficial thrombophlebitis of the target saphenous vein with scarring in the treatment section
6. Pregnant or breastfeeding
7. Known sensitivity or allergic response to Sodium Tetradecyl Sulfate (STS)
8. Known high risk of thrombosis
9. Known history of deep vein thrombus (DVT) or pulmonary embolism (PE), known history of acute superficial vein thrombus, known hypercoagulable condition, post thrombotic syndrome
10. Known history of anaphylaxis or presence of multiple severe allergies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2020-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Meissner, MD, Study Chair — Vascular and Endovascular Surgery Clinic at UWMC
Locations (5):
- United States (5):
  - The Vascular Experts, Darien, Connecticut
  - Capitol Vein and Laser Centers, Frederick, Maryland
  - Southeastern Surgical Associates, Hyannis, Massachusetts
  - Englegwood Hospital and Medical Center, Englewood, New Jersey
  - Lake Washington Vascular, PLLC, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ClariVein RES 1% Injection | ClariVein RES 3% Injection
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ClariVein RES 1% Injection | ClariVein RES 3% Injection | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 19
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 25.6 (4.54) | 27.1 (5.35) | 26.3 (4.86)
Ultrasound Parameters at Screening: Leg Assessed [Count of Participants; unit: Participants]
  Right | 7 | 3 | 10
  Left | 3 | 6 | 9
Retrograde Flow [Count of Participants; unit: Participants] | 10 | 9 | 19
Patient-Reported Symptoms 7-Day Symptom Questionnaire (Average Daily Total Symptom Score [Mean (Standard Deviation); unit: units on a scale] — 7 Day Symptom Questionnaire. Subjects self reported each symptom on a daily basis for 7 consecutive days prior to study day 1. Response to each system was rated on a common 4-point response scale, with lower scores representing better daily health outcomes (4=all day, 3=several times today, 2=once today, 1=not today). Mean is calculated across daily responses for each of the symptoms. Weekly average score was calculated if at least 4 daily scores were present. Daily total symptom score is derived as sum of responses across all symptoms (range 5 to 20). More than 2 items missing, then no score
  units on a scale | 10.6 (3.39) | 11.3 (4.18) | 10.9 (3.76)
Saphenous Vein Reflux [Count of Participants; unit: Participants] — Evaluated by way of duplex ultrasound and read by Core Lab. Elimination of saphenous vein reflux can be achieved when ultrasound images demonstrate vein closure (no discrete open segment of vein > 5cm in length within the treatment section of the selected saphenous vein), or vein competency (defined as absence of retrograde flow > 0.5 seconds within any open portions of the treatment section of the selected saphenous vein) as assessed by duplex ultrasound. Responder = subjects who satisfies criteria for elimination of saphenous vein reflux
  Participants | 10 | 9 | 19
Length of Vein Section to be Treated [Mean (Standard Deviation); unit: centimeters (cm)] | 37.8 (6.49) | 34.6 (15.27) | 36.3 (11.29)
Diameter of Vein Section to be Treated [Mean (Standard Deviation); unit: centimeters (cm)] | 5.41 (0.845) | 9.08 (7.490) | 7.15 (5.369)

OUTCOME MEASURES:

1. Primary Outcome: Patient-Reported Symptoms 7-Day Symptom Questionnaire (Heaviness, Achiness, Swelling, Throbbing & Itching) to Evaluate Improvement in Subject Reported Symptoms.
Description: The VEINES-QOL (VEnous INsufficiency Epidemiological and Economic Study Quality of Life) comprises 25 items that quantify disease effect on quality-of-life, & a symptom questionnaire (VEINES-Sym) with 10 items that measure physical symptoms. A subset of the reported symptoms to Question 1 of the VEINES QOL/Sym is referred to as the 7-Day Symptom Questionnaire was used in this study. Subject response to each symptom was rated on a common 4-point response scale with lower scores representing better daily health outcomes (4=all day, 3=several times today, 2=once today, 1=not today). Weekly average score was calculated if at least 4 daily scores were present in the previous week. Daily total symptom score derived as sum of the responses across all symptoms (range = 5 to 20) Improvement in patient reported symptoms using the 7-Day Symptom Questionnaire (Heaviness, Achiness, Swelling, Throbbing & Itching) at post-treatment Week 12 compared to Baseline is the primary endpoint of this study.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ClariVein RES 1% Injection | ClariVein RES 3% Injection
Number analyzed (Participants) | 10 | 9
units on a scale | 7.2 (3.00) | 6.2 (1.87)
Statistical Analysis 1: Comparison: ClariVein RES 1% Injection vs ClariVein RES 3% Injection; Continuous variables summarized using descriptive statistics, specifically the mean, median, standard deviation, minimum and maximum. Categorical variables summarized using frequencies and percentages. All statistical tests will be performed at the 0.05 significance level (p -value ≤ 0.050) unless otherwise indicated. For efficacy analyses, missing post-treatment data will be imputed using last observation carried forward (LOCF). Missing safety data will not be imputed; Test type: Other — The null hypothesis is that the mean change from baseline for the primary efficacy endpoint=0. The alternative hypothesis is that the mean change does not =0. The primary analysis will be a one-sample t-test for both treatment groups combined, to test the null hypothesis that the mean change from baseline equals 0. Primary analysis will be performed for each treatment group separately; p < 0.001, t-test, 2 sided — This p-value corresponds to the change from Baseline to Week 12 for both treatment groups (ClariVein RES 1% Injection and ClariVein RES 3% Injection) combined; One-Sample; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-6.2 to -2.3]
Statistical Analysis 2: Comparison: ClariVein RES 1% Injection; All statistical tests will be performed at the 0.05 significance level (p -value ≤ 0.050) unless otherwise indicated; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.011, t-test, 2 sided — This p-value corresponds to the change from Baseline to Week 12 for the ClariVein RES 1% Injection treatment group; One-Sample; Mean Difference (Final Values) = -3.4, 95% CI 2-sided [-5.8 to -1.0]
Statistical Analysis 3: Comparison: ClariVein RES 3% Injection; All statistical tests will be performed at the 0.05 significance level (p -value ≤ 0.050) unless otherwise indicated; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.010, t-test, 2 sided — This p-value corresponds to the change from Baseline to Week 12 for the ClariVein RES 3% Injection treatment group; One-Sample; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-8.7 to -1.6]
Statistical Analysis 4: Comparison: ClariVein RES 1% Injection vs ClariVein RES 3% Injection; All statistical tests will be performed at the 0.05 significance level (p -value ≤ 0.050) unless otherwise indicated; Test type: Other — An ANCOVA was performed to compare the change from baseline for ClariVein RES 1% Injection versus ClariVein RES 3% Injection with treatment as the class variable and with baseline score as the covariate; p = 0.531, ANCOVA — This p-value corresponds to the difference between treatment groups (ClariVein RES 1% Injection versus ClariVein RES 3% Injection); Least-Squares Mean Difference = -1.2, 95% CI 2-sided [-3.7 to 1.3]

2. Secondary Outcome: Elimination of Saphenous Vein Reflux
Description: Evaluated by way of duplex ultrasound and read by Core Lab. Elimination of saphenous vein reflux can be achieved when ultrasound images demonstrate vein closure (no discrete open segment of vein > 5cm in length within the treatment section of the selected saphenous vein), or vein competency (defined as absence of retrograde flow > 0.5 seconds within any open portions of the treatment section of the selected saphenous vein) as assessed by duplex ultrasound. Responder = subjects who satisfies criteria for elimination of saphenous vein reflux
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ClariVein RES 1% Injection | ClariVein RES 3% Injection
Number analyzed (Participants) | 10 | 9
Participants
  Vein Closure : Yes | 5 | 9
  Vein Closure : No | 5 | 0
  Vein Closure : Missing | 0 | 0
  Vein Competency : Yes | 2 | 0
  Vein Competency : No | 3 | 0
  Vein Competency : Missing | 0 | 0
  Vein Competency: No open segments > 5cm | 5 | 9
  Saphenous Vein Reflux: Non-Responder | 3 | 0
  Saphenous Vein Reflux: Responder | 7 | 9
Statistical Analysis 1: Comparison: ClariVein RES 1% Injection vs ClariVein RES 3% Injection; The secondary efficacy endpoint, the elimination of saphenous vein reflux at Week 12 posttreatment, will be summarized for both treatments combined using the count and percentage, together with a 95% Wilson (score) confidence interval for the proportion; Test type: Other; Descriptive (Percentage) = 94.4, 95% CI 2-sided [72.7 to 99.9] — The count of the combined treatment group for the elimination of saphenous vein reflux at Week 12 posttreatment is 17/18 (94.4%)
Statistical Analysis 2: Comparison: ClariVein RES 1% Injection vs ClariVein RES 3% Injection; For elimination of saphenous vein reflux at Week 12 posttreatment, the treatment difference for ClariVein RES 1% Injection versus ClariVein RES 3% Injection for the proportion was assessed by a chi-square test together with a 95% Wilson (score) confidence interval for the treatment difference; Test type: Other; p = 1.000, Chi-squared — All statistical tests will be performed at the 0.05 significance level (p -value ≤ 0.050) unless otherwise indicated; Percentage Difference = 11.1, 95% CI 2-sided [-20.5 to 42.8]

ADVERSE EVENTS:
Time Frame: AE data collection began after ICF is signed and continued until completion of subject's Week 12 post-treatment follow-up visit (Visit 6). Any AE or SAE having an onset after the completion of Visit 6 (end of the study visit) was not collected or reported unless the Investigator determined event to be related to the study drug.
Arm/Group | ClariVein RES 1% Injection | ClariVein RES 3% Injection
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 1/10 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ClariVein RES 1% Injection (N=10) | ClariVein RES 3% Injection (N=9)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Blister (From Compression Sock)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 2 (2) — superficial thrombophlebitis.
Infusion Site Bruising (General disorders) | 1 (1) | 1 (1) — Bruising at Access Site

LIMITATIONS AND CAVEATS:
A total of 19 subjects were enrolled in the study. The study was terminated for administrative reasons; there were no safety or efficacy concerns. It was determined by the sponsor that the Phase 3 protocol, which is designed to closely mimic the Phase 2 protocol, would be adequate to collect safety and efficacy assessments with minor adjustments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT03311269/Prot_SAP_000.pdf